CLINICAL TRIAL: NCT06675916
Title: Assessment of PENG Block Analgesia Versus Intra-articular Infiltration in Hip Prosthesis Surgery
Acronym: API
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-A00539-32
Record Dates: First submitted 2024-06-03; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG block (Experimental): Total hip prosthesis with infiltration of lidocaine hydrochloride by ultrasound-guided PENG block
  Interventions: Procedure: PENG Block with lidocaine hydrochloride
- Intra-articular infiltration (Active Comparator): Total hip prosthesis with intra-articular infiltration of lidocaine hydrochloride
  Interventions: Procedure: Intra-articular infiltration with lidocaine hydrochloride

INTERVENTIONS:
Procedure: PENG Block with lidocaine hydrochloride — Intervention is ultrasound-guided PENG block analgesia with lidocaine hydrochloride
  Arms: PENG block
Procedure: Intra-articular infiltration with lidocaine hydrochloride — Intervention is intra-articular analgesia with lidocaine hydrochloride
  Arms: Intra-articular infiltration

SUMMARY:
After hip arthroplasty, pain intensity is maximum within the first 6 hours and is then estimated to last between 36 and 72 hours.

Pain management (analgesia) after hip prosthetic surgery remains a challenge. A bad analgesic treatment can result in delay in mobilization/ambulation and thus increase duration of patient's stay which can have a significant economic impact.

The different recognized analgesia techniques (intra-articular infiltration and peripheral nerve blocks) are effective but have shown certain limits.

A new peripheral nerve block, the PENG block has shown very encouraging results on postoperative analgesia quality.

In this context, this research is based on the hypothesis that ultrasound-guided PENG block could provide more effective analgesia than intra-articular infiltration during mini-invasive anterior hip prosthesis surgery.

DETAILED DESCRIPTION:
Each year, around140 000 patients undergo total hip arthroplasty. After hip arthroplasty, pain intensity is maximum within the first 6 hours and is then estimated to last between 36 and 72 hours. However, more and more patients want to no longer suffer after surgery. Indeed, if postoperative pain is moderate at rest, it is often exacerbated by movement. Severe pain occurs in 50 % of patients at rest and in 70% of patients during mobilization.

Pain management (analgesia) after hip prosthetic surgery remains a challenge for the anesthesiologist. A bad analgesic treatment can result in delay in mobilization/ambulation and thus increase duration of patient's stay which can have a significant economic impact. Quality analgesia is therefore essential to reduce post-operative pain and improve functional rehabilitation in patients undergoing hip surgery.

The different recognized analgesia techniques (intra-articular infiltration and peripheral nerve blocks) are effective but have shown certain limits: rapid and non-lasting effect of analgesia or poor targeting of all nerves of hip joint.

A new peripheral nerve block, the PENG block, identified during a recent anatomical study in 2018, has shown very encouraging results on postoperative analgesia quality on several small series of patients.

In this context, this research is based on the hypothesis that ultrasound-guided PENG block could provide more effective analgesia than intra-articular infiltration and therefore reduce the intraoperative opioid consumption during mini-invasive anterior hip prosthesis surgery under general anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, over 18 years old.
* Patient scheduled for hip prosthesis placement via the anterior approach

Exclusion Criteria:

* Patient with local anesthesia contraindication.
* Patient with a high level of dependency, defined by level 1 or 2 of Iso Ressources Group (GIR).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Morphine dose | 1 day
  Primary outcome measure is the total morphine quantity administered intraoperatively, in milligrams

SECONDARY OUTCOMES:
Pain level | Day 0, 1, 7 and 45
  Pain is assessed with Visual Analogic Scale (0 - 10 points). 0 is the lowest pain value (patient has no pain) whereas 10 is the highest pain value.
Patient quality of life | Day 1, 7 and 45
  Quality of life is assessed with EQ-5D-5L (EUROQOL - 5 dimensions - 5 levels) questionnaire (0 - 100 points). 0 means the worst quality of life whereas 100 means the best quality of life.
Hip symptoms and limitations | Day 45
  Hip symptoms and limitations assessment relies on HOOS questionnaire (0 - 100 points). 0 is the worst possible score whereas 100 is the best possible score (no symptoms and no limitations)
Hip impact on daily life | Day 45
  Hip impact on daily life is assessed with OXFORD questionnaire (12 - 60 points). 12 is the best patient score (hip has no impact on patient daily life) whereas 60 is the worst patient score

CONTACTS AND LOCATIONS:
Locations (1):
- Médipôle Hôpital Privé, Villeurbanne, France

IPD SHARING:
Plan to Share IPD: No